CLINICAL TRIAL: NCT01321840
Title: Investigation of Cortical Plasticity in a Complex Intervention for Endometriosis
Brief Title: Cortical Plasticity in a Complex Intervention for Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Florian Beissner, Dr. phil. nat., University of Jena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Jena-Endo-01
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; pain; sart; autonomic nervous system; fMRI; perfusion; connectivity; hypnotherapy; traditional Chinese medicine
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): This group will be treated with SART.
  Interventions: Procedure: Specific Autoregulation Therapy (SART)
- No treatment (No Intervention): This group will not be treated with SART but will regularly be examined by a gynecologist to detect sudden aggravation of the disease.

INTERVENTIONS:
Procedure: Specific Autoregulation Therapy (SART) — Complex intervention involving acupuncture and hypnotherapeutic techniques after an extensive diagnosis using chinese medical concepts. Patients will receive a maximum of 10 treatments, which are delivered weekly.
  Arms: Treatment

SUMMARY:
The aim of the study is to test, if patients suffering from Endometriosis show changes in their brain function, when being treated with SART (Systemic Autoregulation Therapy), a complex intervention consisting of interventions from Traditional Chinese Medicine (TCM) and Western Hypnotherapy. Functional and structural brain changes are assessed using Magnetic Resonance Imaging data which are analyzed by means of voxel-based morphometry (VBM), connectivity and perfusion analysis. A third outcome measure are changes of patients' heart rate variability, indicating the activity of their autonomic nervous system.

With a number of questionnaires, changes in dysmenorrhea, chronic pelvic pain, menstruation regularity, dyspareunia, defecation pain, and quality of life are assessed during the SART treatment.

During the treatment, we expect to see changes in cortical thickness, functional connectivity and perfusion of pain-related areas of the cortex, that correlate with the changes in heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* clinically or histologically ensured diagnosis of Endometriosis
* preoperative and postoperative recurring ailments related to Endometriosis
* no hormone therapy (GnRH analogues, contraceptives)
* sufficient understanding of the German or English language
* persisting pain during menstruation (also in between)
* voluntary participation after information on the possible benefits and risks of the examination and intervention
* written informed consent

Exclusion Criteria:

* alcohol addiction, drug addiction
* pregnancy
* diseases and other criteria, preventing an MRI examination:
* pacemaker
* neurostimulator or drug pump
* metal parts in the body (implants, splinters, etc.)
* claustrophobia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Brain function | 12 weeks
  Changes in cortical thickness, functional connectivity and perfusion of brain areas related to the processing of pain and emotions.

SECONDARY OUTCOMES:
Reduction of pain | 12 weeks
  Reduction of pain by 50% or more (dichotomous).
Pain scores | 12 wks
  Changes (ordinal) in pain scores as assessed by the questionnaire of the German Society For The Study Of Pain (DGSS).
Quality of life | 12 wks
  Changes (ordinal) in the quality of life score as assessed by the questionnaire of the German Society For The Study Of Pain (DGSS).
Endometriosis-related symptoms | 12 wks
  Normalization of menstruation, pelvic pain, dyspareunia, defecation pain as assessed by the Erlangen Endometriosis questionnaire.
HRV (HF, LF, LF/HF) | 12 wks
  heart rate variability parameters

CONTACTS AND LOCATIONS:
Overall Officials: Florian Beissner, Dr.phil.nat., Study Director — Pain & Autonomics - Integrative Research, Klinik für Psychiatrie und Psychotherapie, Jena
Locations (2):
- Germany (2):
  - Pain & Autonomics - Integrative Research, Klinik für Psychiatrie und Psychotherapie, Jena
  - Frauenklinik der Technischen Universität München, München

REFERENCES:
- [Result] Meissner K, Schweizer-Arau A, Limmer A, Preibisch C, Popovici RM, Lange I, de Oriol B, Beissner F. Psychotherapy With Somatosensory Stimulation for Endometriosis-Associated Pain: A Randomized Controlled Trial. Obstet Gynecol. 2016 Nov;128(5):1134-1142. doi: 10.1097/AOG.0000000000001691. PMID 27741200
- [Derived] Beissner F, Preibisch C, Schweizer-Arau A, Popovici RM, Meissner K. Psychotherapy With Somatosensory Stimulation for Endometriosis-Associated Pain: The Role of the Anterior Hippocampus. Biol Psychiatry. 2018 Nov 15;84(10):734-742. doi: 10.1016/j.biopsych.2017.01.006. Epub 2017 Jan 16. PMID 28258747